CLINICAL TRIAL: NCT05247060
Title: Orthostatic Hypotension in Hypertensive Patient Hospitalized in Internal Medicine - Prevalence, Concomitant Conditions and Outcomes
Brief Title: Orthostatic Hypotension in Hypertensive Patient Hospitalized in Internal Medicine
Acronym: IP-OP
Status: Completed | Type: Observational
Sponsor: Fadoi Foundation, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: FADOI.02.2018
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hospitalization
Keywords: orthostatic hypotension; Internal Medicine
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertensive Patients Hospitalized in Internal Medicine: Clinical data will be collected from all consecutive patients diagnosed with arterial hypertension hospitalized in Internal Medicine and able to assume the erect station
  Interventions: Other: no experimental intervention

INTERVENTIONS:
Other: no experimental intervention — There will not be any experimental intervention. The study will be conducted according with normal clinical practice

SUMMARY:
The two scientific societies FADOI and SIIA have decided to start a collaborative study protocol that, through the application of a simple and homogeneous method to diagnose orthostatic hypotension, aims to estimate prevalence, conditions associates and outcomes in a cohort of patients admitted to Internal Medicine Departments and with known or newly diagnosed arterial hypertension.

DETAILED DESCRIPTION:
The IP-OP study, is an observational, multicenter, prospective, national study that provides for the involvement of 34 Operating Units of Internal Medicine, and the recording of data relating to 1000 hospitalized adults.

The clinical data of all consecutive patients diagnosed with arterial hypertension hospitalized in Internal Medicine and able to take the erect station will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presence of arterial hypertension (known or discovered at hospitalization)
* Signature of Informed Consent

Exclusion Criteria:

* Patients unable to take the standing station for a few minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients diagnosed with arterial hypertension hospitalized in Internal Medicine and able to assume the erect station
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
clinical conditions ( physiological parameters, copatologies) associated with the presence of orthostatic hypotension | 4 months
  Identification, through a multivariate analysis, of the clinical conditions associated with the presence of orthostatic hypotension in the population of hypertensive patients admitted to Internal Medicine

SECONDARY OUTCOMES:
Prevalence of orthostatic hypotension | 4 months
  Prevalence of orthostatic hypotension among hypertensive patients admitted to Internal Medicine
Gender differences in prevalence and conditions associated with orthostatic hypotension | 4 months
  Assessment of possible gender differences in prevalence and conditions associated with orthostatic hypotension
Level of cognitive impairment of the subjects studied, and relationship with orthostatic hypotension | 4 months
  Evaluation in the initial visit of the level of cognitive impairment of the subjects studied, and relationship with orthostatic hypotension
Relationship between orthostatic hypotension and a Fragility Index | 4 months
  Evaluation of the relationship between orthostatic hypotension and a Fragility Index
Relationship between orthostatic hypotension and comorbidity by calculating the index of Charlson comorbidity | 4 months
  Evaluation of the relationship between orthostatic hypotension and comorbidity by calculating the index of Charlson comorbidity
Prescription drugs on the presence and severity of hypotension Orthostatic | 4 months
  Analysis of the impact of prescription drugs on the presence and severity of hypotension Orthostatic
Presence of orthostatic hypertension | 4 months
  Evaluation of the presence of orthostatic hypertension
After 6-12-24-36 months from the index hospitalization, of the state of health of all the subjects evaluated | 6-12-24-36 months from hospitalization
  Evaluation, after 6-12-24-36 months from the index hospitalization, of the state of health of all the subjects evaluated, reporting the possible onset of falls, major cardiovascular events (stroke, TIA, myocardial infarction, arrhythmias) or death.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Fontanella, MD, Study Director — FADOI FOUNDATION
Locations (33):
- Italy (33):
  - Ospedale Civile, Legnano, (MI)
  - Ospedale "S. Maria", Borgo Val di Taro, (PR)
  - Ospedale Luini Confalonieri, Luino, (VA)
  - P.O. di Rete Bassano, Bassano del Grappa, (VI)
  - P.O. "SS. Filippo e Nicola", Avezzano, AQ
  - Ospedale Civ. "S. Maria Incoronata dell'Olmo", Cava de' Tirreni, SA
  - Ospedale Maggiore, Chieri, TO
  - Ospedale di Sant'Agata dei Goti, Benevento
  - Ospedali Civili di Brescia, Brescia
  - AO Sant'Anna e San Sebastiano, Caserta
  - Ospedale ARNAS Garibaldi, Catania
  - Ospedale Sant'Anna, Como
  - Ospedale di Ceva, Cuneo
  - AOU Careggi, Florence
  - Ospedale di Galliera, Genova
  - Ospedale San Salvatore, L’Aquila
  - Ospedale Niguarda, Milan
  - Ospedale San Luca, Milan
  - Ospedale Buon Consiglio Fatebenefratelli, Napoli
  - Ospedale Cardarelli, Napoli
  - Ospedale di Piove di Sacco, Padua
  - Ospedale San Jacopo, Pistoia
  - P.O. "S. Maria delle Grazie", Pozzuoli
  - Ospedale Fatebenefratelli, Roma
  - Ospedale Santa Maria della Misericordia, Rovigo
  - AOU San Giovanni di Dio e Ruggi d'Aragona, Salerno
  - Ospedale Abbadia San Salvatore, Siena
  - PO "Umberto I", Syracuse
  - Ospedale "Città della Salute", Torino
  - Ospedale Cà Foncello, Treviso
  - Ospedale di Circolo, Varese
  - AOUI - Borgo Trento, Verona
  - Ospedale Versilia, Viareggio

IPD SHARING:
Plan to Share IPD: No